CLINICAL TRIAL: NCT03987061
Title: Physician-initiated Trial Investigating the MOTIV™ Bioresorbable Scaffold (Reva Medical) for the Treatment of Below-The-Knee Artery Disease
Brief Title: MOTIV Bioresorbable Scaffold in BTK Artery Disease
Acronym: MOTIV BVS BTK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Sabrina Overhagen (Other)
Responsible Party: Sponsor-Investigator, Dr. Sabrina Overhagen, Director, FCRE (Foundation for Cardiovascular Research and Education)
Organization: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCRE-190131
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Application of the MOTIV Bioresorbable Scaffold in Patients with Lesions Below-The-Knee (BTK)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOTIV bioresorbable vascular scaffold (Experimental): MOTIV bioresorbable vascular scaffold for below-the-knee artery disease
  Interventions: Device: MOTIV BVS

INTERVENTIONS:
Device: MOTIV BVS — MOTIVS BVS in below-the-knee artery disease

SUMMARY:
The objective of this clinical evaluation is to evaluate the immediate and long-term (up to 36 months) outcome of the MOTIV™ Bioresorbable Scaffold (Reva Medical) in a controlled prospective investigation for the treatment of patients with rest pain or minor tissue loss (CLI) due to the presence of lesions of max 100mm in length at the level of the below-the-knee arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient presenting with rest pain or minor tissue loss (Rutherford classification from 4 to 5)
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrollment in the study - Patient has a projected life-expectancy of at least 24-months
* Patient is eligible for treatment with the MOTIV™ Bioresorbable Scaffold
* Male, infertile female, or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure
* De novo lesion or Restenotic lesion after PTA in the infrapopliteal arteries, suitable for endovascular therapy
* Target vessel diameter visually estimated to be ≥2.5mm and ≤3.50mm
* Guidewire and delivery system successfully traversed the lesion
* Total target lesion is maximally 100mm
* Definition of Target Lesion is:

  1. short de novo or Restenotic lesion after PTA or
  2. a short residual flow-limiting dissection or restenosis after PTA of a longer lesion

Exclusion Criteria:

* The reference segment diameter is not suitable for the available stent design
* Untreated flow-limiting aortoiliac stenotic disease
* Perioperative unsuccessful ipsilateral percutaneous vascular procedure to treat inflow disease just prior to enrollment.
* Any previous surgery in the target vessel
* Aneurysm located at the target vessel
* Non-atherosclerothic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* Severe medical comorbidities (untreated CAD/CHF, severe COPD, metastatic malignancy, dementia, etc) or other medical condition that would preclude compliance with the study protocol or 2-year life expectancy.
* Major distal amputation (above the transmetatarsal) in the study or non-study limb.
* Septicemia or bacteremia
* Any previously known coagulation disorder, including hypercoagulability
* Contraindication to anticoagulation or antiplatelet therapy
* Known allergies to scaffold or scaffold components
* Known allergies to contrast media that cannot be adequately premedicated prior to the study procedure
* Patient with known hypersensitivity to heparin-induced thrombocytopenia (HIT) type II
* Currently participating in another clinical research trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
efficacy endpoint - Primary Patency rate at 12-months post-op | 12 months post-op
  Primary patency defined as no evidence of at least 50% restenosis or reocclusion within the originally treated lesion based on color-flow-duplex ultrasound (CFDU) measuring a peak systolic velocity ratio ≤2.5, and/or angiography (left at the discretion of the investigator) without target lesion revascularization (TLR) within 12 months.
safety endpoint - rate of serious device-related adverse events within 30 days post-op | 30 days post-op
  Proportion of subjects who experience serious device-related adverse events within 30 days post-procedure.

SECONDARY OUTCOMES:
Technical Success | 1-day post-op
  Technical Success, defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30%
Primary Patency rate at follow-up visits | 1 month, 6 months, 12 months, 24 months and 36 months post-op
  Primary patency rate defined as no evidence of at least 50% restenosis or reocclusion within the originally treated lesion based on color-flow-duplex ultrasound (CFDU) measuring a peak systolic velocity ratio ≤2.5, and/or angiography (left at the discretion of the investigator) without target lesion revascularization (TLR) within 12 months.
Clinically-driven target lesion revascularization (TLR) at 1, 6, 12, 24 and 36-months | 1 month, 6 months, 12 months, 24 months and 36 months post-op
  Clinically-driven (drop in 1 Rutherford Classification) target lesion revascularization (TLR) is defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the device/PTA edge
Limb-Salvage rate at follow-up visits | 1 month, 6 months, 12 months, 24 months and 36 months post-op
  Major amputation is defined as amputation at or above the ankle, as opposed to minor amputation, being an amputation at or below metatarsal level, preserving functionality of the foot.
Clinical success at follow-up visits | 1 day post-op and 1 month, 6 months, 12 months, 24 months and 36 months post-op
  Clinical success at follow-up is defined as an improvement of Rutherford classification at 1 day and 1-, 6-, 12-, 24- and 36-months follow-up of one class or more as compared to the pre-procedural Rutherford Classification.
Serious adverse events during the study (within 36 months post-op) | within 36 months post-op
  Serious adverse events as defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Torsello, Prof. Dr., Study Director — Foundation for Cardiovascular Research and Education
Locations (8):
- Hospital Floridsdorf, Vienna, Austria
- Germany (7):
  - Klinikum Hochsauerland, Arnsberg
  - Bad Oeyhausen Klinik für Allgemeine und Interventionelle Kardiologie/Angiologie, Bad Oeynhausen
  - Medizinische Versorgungszentren GmbH, Berlin
  - University Hospital Leipzig, Angiology, Leipzig
  - Katholisches Klinikum Mainz; Akademisches Lehrkrankenhaus der Johannes Gutenberg-Universität Mainz, Mainz
  - St. Franziskus-Hospital, Münster
  - University Hospital Münster, Angiology, Münster

IPD SHARING:
Plan to Share IPD: No